CLINICAL TRIAL: NCT04373707
Title: Effectiveness of Weight-adjusted Prophylactic Low Molecular Weight Heparin Doses Compared With Lower Fixed Prophylactic Doses to Prevent Venous Thromboembolism in COVID-2019. The Multicenter Randomized Controlled Open-label Trial COVI-DOSE
Brief Title: Weight-Adjusted vs Fixed Low Doses of Low Molecular Weight Heparin For Venous Thromboembolism Prevention in COVID-19
Acronym: COVI-DOSE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Ministry of Health, France (Other Government); Grand Est Region (Unknown); University Hospital of Saint-Etienne (Other)
Responsible Party: Principal Investigator, Stéphane Zuily, MD, PhD, Central Hospital, Nancy, France
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-001709-21
Record Dates: First submitted 2020-05-01; First posted 2020-05-04 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: COVID; Thrombosis; Pulmonary Embolism; Deep Vein Thrombosis
Keywords: COVID; Thrombosis; Venous Thromboembolism; Pulmonary Embolism; Deep Vein Thrombosis; Low Molecular Weight Heparin
MeSH Terms: conditions — Thrombosis; Pulmonary Embolism; Venous Thrombosis; Venous Thromboembolism | interventions — Enoxaparin; Tinzaparin; Nadroparin; Dalteparin

STUDY DESIGN:
Intervention Model Description: Multicenter randomized (1:1) controlled open-label trial, stratified on disease severity (admission to ICU or not)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low Prophylactic Dose of Low Molecular Weight Heparin (Active Comparator): Enoxaparin, Tinzaparin, Nadroparin, Dalteparin
  Interventions: Drug: Enoxaparin
- Weight-Adjusted Prophylactic Dose Low Molecular Weight Heparin (Experimental): Enoxaparin, Tinzaparin, Nadroparin, Dalteparin
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin — For example (Enoxaparin):
  * 4000IU twice a day in patients <50kg
  * 5000IU twice a day in patients 50-70kg
  * 6000IU twice a day in patients 70-100kg
  * 7000IU twice a day in patients above 100kg
  Other Names: Tinzaparin; Nadroparin; Dalteparin
  Arms: Weight-Adjusted Prophylactic Dose Low Molecular Weight Heparin
Drug: Enoxaparin — For example (Enoxaparin): From 4000IU once a day in patients admitted in medical ward to 4000IU twice a day in patients admitted in the ICU. In patients with severe renal insufficiency (GFR=15-30 mL/min/1.73m²), LMWH doses will be reduced by 50%.
  Other Names: Tinzaparin; Nadroparin; Dalteparin
  Arms: Low Prophylactic Dose of Low Molecular Weight Heparin

SUMMARY:
Worldwide observational studies indicate a significant prothrombogenic effect associated with SARS-CoV-2 infection with a high incidence of venous thromboembolism (VTE), notably life-threatening pulmonary embolism.

According to recommendations for acute medical illnesses, all COVID-19 hospitalized patients should be given VTE prophylaxis such as a low molecular weight heparin (LMWH). A standard prophylactic dose (eg. Enoxaparin 4000IU once daily) could be insufficient in obese patients and VTE has been reported in patients treated with a standard prophylactic dose.

In COVID-19 patients, guidelines from several international societies confirm the existence of an hypercoagulability and the importance of thromboprophylaxis but the "optimal dose is unknown" and comparative studies are needed.

In view of these elements, carrying out a trial comparing various therapeutic strategies for the prevention of VTE in hospitalized patients with COVID-19 constitutes a health emergency.

Thus, we hypothesize that an increased prophylactic dose of weight-adjusted LMWH would be greater than a lower prophylactic dose of LMWH to reduce the risk of life-threatening VTE in hospitalized patients. The benefit-risk balance of this increase dose will be carefully evaluated because of bleeding complications favored by possible renal / hepatic dysfunctions, drug interactions or invasive procedures in COVID-19 patients.

This multicenter randomized (1:1) open-label controlled trial will randomize hospitalized adults with COVID-19 infection to weight-adjusted prophylactic dose vs. lower prophylactic dose of LMWH.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient hospitalized for a probable/confirmed COVID-19 infection (confirmed by serology/polymerase chain reaction or by radiologic signs of COVID-19 pneumonia in the setting of clinical and laboratory abnormalities suggestive of a SARS-CoV-2 infection)
* Signed informed consent
* Patient affiliated to the Social Security

Exclusion Criteria:

* Renal insufficiency with a GFR<15 mL/min/1.73m²
* Acute kidney injury KDIGO3
* Prophylactic dose of low molecular weight heparin for more than 3 days
* Curative dose of low molecular weight heparin for more than 1 day
* Recurrent catheter/hemodialysis access thromboses
* ECMO required in the next 24h
* Contraindication to low molecular weight heparin
* High bleeding risk (e.g. uncontrolled severe systemic hypertension, recent major bleeding, disseminated intravascular coagulopathy, thrombocytopenia < 75G/L)
* History of heparin-induced thrombocytopenia
* Contraindication to blood-derived products
* Impossibility to perform a doppler ultrasound of the lower limbs (e.g. above the knee amputation, severe burn injuries)
* Expected death in the next 48h
* Vulnerable subjects according to articles L. 1121-5, L. 1121-7 et L1121-8 of French Public Health Code

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-09-14 (Actual)

PRIMARY OUTCOMES:
Venous thromboembolism | hospitalization stay (up to 28 days)
  Risk of deep vein thrombosis or pulmonary embolism or venous thromboembolism-related death

SECONDARY OUTCOMES:
Major bleeding | hospitalization stay (up to 28 days)
  Risk of major bleeding defined by the ISTH
Major Bleeding and Clinically Relevant Non-Major Bleeding | hospitalization stay (up to 28 days)
  Risk of Major Bleeding and Clinically Relevant Non-Major Bleeding Defined by the ISTH
Net Clinical Benefit | hospitalization stay (up to 28 days) and 60 days
  Risk of Venous Thromboembolism and Major Bleeding
Venous Thromboembolism at other sites | hospitalization stay (up to 28 days)
  Risk of venous thrombosis at other sites: e.g. superficial vein, catheters, hemodialysis access, ECMO, splanchnic, encephalic, upper limb
Arterial Thrombosis | hospitalization stay (up to 28 days)
  Risk of arterial thrombosis at any sites
All-Cause Mortality | hospitalization stay (up to 28 days) and 60 days
  Risk of all-cause mortality
Factors associated with the risk of venous thromboembolism | hospitalization stay (up to 28 days)
  Identification of associations between the risk of venous thromboembolism and clinical (eg. past medical history of thrombosis, cardiovascular risk factors, treatments, severity of COVID-19) and laboratory variables (e.g. D-dimers, fibrinogen, CRP) collected in the eCRF

CONTACTS AND LOCATIONS:
Overall Officials: El Mehdi Siaghy, Study Director — Research and Innovation Department, Nancy University Hospital; Stéphane Zuily, MD, PhD, Principal Investigator — Nancy Academic Hospital
Locations (17):
- France (17):
  - Amiens Academic Hospital, Amiens
  - Besançon Academic Hospital, Besançon
  - Brest Academic Hospital, Brest
  - Civil Hospital, Colmar
  - Dijon Academic Hospital, Dijon
  - Kremlin Bicêtre Academic Hospital, Le Kremlin-Bicêtre
  - Lille Academic Hospital, Lille
  - Groupe Hospitalier Unéos, Metz
  - Metz-Thionville Regional Hospital, Metz
  - Montpellier Academic Hospital, Montpellier
  - Emile Muller Hospital, Mulhouse
  - Nancy Academic Hospital, Nancy
  - George Pompidou European Hospital, Paris
  - Lariboisière Academic Hospital, Paris
  - St Etienne Academic Hospital, Saint-Etienne
  - Strasbourg Academic Hospital, Strasbourg
  - Toulouse Academic Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zuily S, Lefevre B, Sanchez O, Empis de Vendin O, de Ciancio G, Arlet JB, Khider L, Terriat B, Greigert H, Robert CS, Louis G, Trinh-Duc A, Rispal P, Accassat S, Thiery G, Montani D, Azarian R, Meneveau N, Soudet S, Le Mao R, Maurier F, Le Moing V, Quere I, Yelnik CM, Lefebvre N, Martinot M, Delrue M, Benhamou Y, Parent F, Roy PM, Presles E, Goehringer F, Mismetti P, Bertoletti L, Rossignol P, Couturaud F, Wahl D, Thilly N, Laporte S; COVI-DOSE investigators. Effect of weight-adjusted intermediate-dose versus fixed-dose prophylactic anticoagulation with low-molecular-weight heparin on venous thromboembolism among noncritically and critically ill patients with COVID-19: the COVI-DOSE trial, a multicenter, randomised, open-label, phase 4 trial. EClinicalMedicine. 2023 Jun;60:102031. doi: 10.1016/j.eclinm.2023.102031. Epub 2023 Jun 9. PMID 37350990
- [Derived] Flumignan RL, Civile VT, Tinoco JDS, Pascoal PI, Areias LL, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2022 Mar 4;3(3):CD013739. doi: 10.1002/14651858.CD013739.pub2. PMID 35244208
- [Derived] Flumignan RL, Tinoco JDS, Pascoal PI, Areias LL, Cossi MS, Fernandes MI, Costa IK, Souza L, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Prophylactic anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD013739. doi: 10.1002/14651858.CD013739. PMID 33502773
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37350990/